CLINICAL TRIAL: NCT05681013
Title: The Effect of Laughter Therapy on the General Health Status, Sleep Quality, and Stress Level of Nursing Students
Brief Title: The Effect of Laughter Therapy on Nursing Students
Acronym: Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Elif Uner, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 739904
Record Dates: First submitted 2022-12-11; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Mental Stress; Insomnia; Sleep Disorder; Mental Health Disorder
Keywords: Sleep Quality; Psychological Stress; General Health; Nursing Students; Laughter Therapy
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Mental Disorders | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Therapy Group (Experimental): A pre-test was administered to all students. In the pre-test application, the Descriptive Information Form, General Health Questionnaire-28, Pittsburgh Sleep Quality Index and Perceived Stress Scale were applied. Experimental and control groups were formed randomly among the students who filled all the scales. Communication groups were established for the students in both groups without being told which group they belonged to. Considering the hours suitable for the experimental group, 8 sessions of laughter therapy were applied for an average of 45 minutes. At the end of the therapy in the last session, a post-test was administered to all of the students. In the post-test application, the Descriptive Information Form, General Health Questionnaire-28, Pittsburgh Sleep Quality Index, and Perceived Stress Scale were applied.
  Interventions: Behavioral: Laughter Therapy
- Control Group (No Intervention): In the pre-test application, the Descriptive Information Form, General Health Questionnaire-28, Pittsburgh Sleep Quality Index, and Perceived Stress Scale were applied. At the end of the therapy in the last session, a post-test was administered to all students. In the post-test application, the Descriptive Information Form, General Health Questionnaire-28, Pittsburgh Sleep Quality Index, and Perceived Stress Scale were applied.

INTERVENTIONS:
Behavioral: Laughter Therapy — The effect of the Laughter Therapy on nursing students
  Arms: Laughter Therapy Group

SUMMARY:
The aim of this study is to determine the effect of laughter therapy on the general health status, sleep quality, and stress level of nursing students.

DETAILED DESCRIPTION:
H1.1: Students who receive laughter therapy will have lower mean scores in the general health questionnaire than students who do not receive laughter therapy.

H1.2: Students who receive laughter therapy will have a lower Pittsburgh sleep quality index score than students who do not receive laughter therapy.

H1.3: Students who receive laughter therapy will have a lower mean stress level than students who do not receive laughter therapy.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Being a 1st or 2nd-year student in the Faculty of Health Sciences, Department of Nursing
* Not have any health problems that may create a communication barrier
* Being in a quiet environment to participate in the online study due to the pandemic period
* Have an internet connection to attend online sessions

Exclusion Criteria:

* Having undergone abdominal surgery in the past three months
* Having a disability to attend regular sessions

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 2 minutes
  It was prepared by the researchers in line with the literature in order to collect data about the individual characteristics of the participants. Form; family structure, gender, income status, marital status, health status, age, etc. It consists of 13 items (pretest-posttest design was applied).
General Health Questionnaire-28 (GHQ-28) | 5 minutes
  It was prepared to detect mental health problems. Individuals who score below 5 on the scale are evaluated as "normal", while individuals who score 5 and above are considered as a "risk group" in terms of mental health (pretest-posttest design was applied).
Pittsburgh Sleep Quality Index (PUKI) | 5 minutes
  "Poor sleep quality" is expressed for individuals who score 5 and above from the scale. The scale consists of 24 items that evaluate sleep quality and disorders by scoring over a one-month period (pretest-posttest design was applied).
Perceived Stress Scale (PSS) | 3 minutes
  The scale, which was prepared to evaluate the perceived stress level of the individual, consists of 14 items. High scores obtained from the scale indicate that the person has a high perception of stress(pretest-posttest design was applied).

CONTACTS AND LOCATIONS:
Overall Officials: Elif Uner, Dr, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No